CLINICAL TRIAL: NCT07376954
Title: Management of Skeletal Class III Malocclusion With Digital Bonded Reverse Twin Block in Mixed Dentition
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Eman Abdelkhabir
Record Dates: First submitted 2025-12-23; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-05

CONDITIONS: Skeletal Class III Malocclusion
Keywords: Skeletal class III malocclusion; Digital bonded reverse twin block; Mixed dentition

STUDY DESIGN:
Intervention Model Description: Digital Bonded Reverse Twin Block
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growing patients with mild skeletal class III (Active Comparator): Digital Bonded Reverse Twin Block
  Interventions: Device: Digital Bonded Reverse Twin Block
- Retrospective skeletal class III patients (No Intervention): Untreated

INTERVENTIONS:
Device: Digital Bonded Reverse Twin Block — Appliance construction:
  * upper blocks (right and left) to be bonded on the anterior region of the maxillary arch.
  * lower blocks (right and left) to be bonded on the posterior region of the mandibular arch.
  Both upper and lower blocks will be produced using Poly-Methyl-Meth-Acrylate (PMMA).
  Upper and lower blocks will interact with each other through coherent specifically designed 70° inclined planes.
  Transparent Polyethylene 0.8mm trays will be used to assist the clinician during the blocks bonding procedures.
  Arms: Growing patients with mild skeletal class III

SUMMARY:
The purpose of this study is to evaluate dentoalveolar & skeletal effects of digital bonded reverse twin block in treatment of skeletal class III malocclusion in mixed dentition.

Class III malocclusion presents significant management and prognostic challenges due to the complex interplay of factors in its etiology. Early diagnosis, planning of adequate therapeutic time and choice of devices to correct malocclusion are the essential keys to successful management of class III in all its forms. Functional appliances are commonly used for the treatment of skeletal class III malocclusion. The aim of this study is to evaluate dentoalveolar & skeletal effects of digital bonded reverse twin block (DBRTB) in treatment of skeletal class III malocclusion in mixed dentition. The digital workflow allows full appliance customization creating a perfect adaptation of the four blocks with patient dental anatomy thus optimizing bonding procedures and block retention. The DBRTB will be designed as four occlusal blocks, two blocks for the upper arch, and two blocks for the lower arch. The upper blocks will be bonded to the anterior part of the maxillary arch, the lower blocks will be bonded to the posterior part of the mandibular arch. Upper and lower blocks will interact with each other through coherent specifically designed 70° inclined planes. Transfer transparent trays will be used to support the bonding procedure of the blocks. Oral Health Related Quality of Life (OHRQoL) assessments will be incorporated as an outcome measure in addressing and measuring clinically meaningful change.

DETAILED DESCRIPTION:
The study includes two groups: (Study design: non-randomized clinical trial)

1. Group 1: control group untreated retrospective data of skeletal class III patients
2. Group 2: patients treated with digital bonded reverse twin block (DBRTB) -Twenty one patients with mild skeletal class III were selected according to specific inclusion criteria and included in the study, these patients were treated with Digital Bonded Reverse Twin Block (DBRTB) to evaluate its dentoalveolar and skeletal effect

Bite registration:

The patient intraoral scan will be obtained using Medit i-700 intraoral scanner. The intraoral scan will be performed according to the constructor's instructions. The software interface of the intra-oral scanner allows the registration of two different maxillo-mandibular relationships (MMRs).

The first MMR scan will be registered in maximum intercuspation occlusion. The second scan will be registered in planned mandibular retrusion for DBRTB design.

Bite registration will be done with the mandible in the most retruded position with an inter- incisal clearance of 2 mm and a clearance of 6 mm in the posterior segment.

To obtain an optimal and reproducible MMR scan in mandibular retrusion, curable resin will be used as a bite registration material.

Two pieces of resin will be used as bite registration material, placing them (one piece per each side of the dentition) onto the occlusal surface of the posterior dentition. Then mandible will be guided in the most retruded position, this will be performed with a brief preliminary patient training. When the mandible reaches the desired backward position, the occlusal resin will be cured on both sides.

Then the two registration pieces of resin will be fully cured outside of the mouth. Once fully polymerized they will be checked for integrity, and they will be placed in occlusion to check that final mandibular retrusion is adequate and conforms to planned retrusion.

Subsequently, patient maxillo-mandibular relationship in mandibular retrusion will be scanned.

During MMR scan acquisition on the right side, only the left piece of resin will be used to maintain mandibular retrusion. Conversely, during MMR scan acquisition on the left side, only the right piece of resin will be used.

At the end of the MMR acquisition process, the software will be able to reorient the maxillary and mandibular scan according to the MMR.

Appliance construction:

The first step of the appliance design is to transform the intra-oral scans into two working models for appliance construction: upper working model and the lower working model.

The DBRTB will be designed as four occlusal bites. Two bites for the upper arch, and two bites for the lower arch. The upper bites will be bonded in the anterior region of the maxillary arch, the lower bites will be bonded in the posterior part of the mandibular arch. Upper and lower bites will interact with each other through coherent specifically designed 70° inclined planes.

After the design process, the following 3D models will be exported as files with STL extension and produced with different procedures and specific purposes:

* upper blocks (right and left) to be bonded on the anterior region of the maxillary arch.
* lower blocks (right and left) to be bonded on the posterior region of the mandibular arch.

Both upper and lower blocks will be produced using Poly-Methyl-Meth-Acrylate (PMMA).

Transparent Polyethylene 0.8mm trays will be used to assist the clinician during the blocks bonding procedures.

Clinical application:

The blocks will be placed inside the transfer transparent trays to ensure a precise bonding position and to reduce the risk of saliva contamination during the bonding procedure.

Intra-oral bonding procedure will be started with the etching of the occlusal surface of the maxillary and mandibular dentition with (Meta Etchant) for 15-20 seconds. Etched dental surfaces will be washed and dried with chair air-flow and light-cured dental adhesive (ORTHOSOLO from Ormco) will be applied to the conditioned dental surfaces. Air-flow will be used again to uniformly spread the adhesive on the teeth surfaces and finally the adhesive will be polymerized for 5 seconds.

BracePaste® Band and Build LC (from American Orthodontics) will be used to bond the blocks. It is decided to use this material to have possibility to distinguish it during blocks debonding.

The bonding material will be placed on the four blocks preliminary positioned into the thermoplastic trays. Subsequently, blocks will be positioned on the dentition with the support of thermoplastic trays and immediately polymerized through the clear trays for 60 seconds per block.

Additionally, the bonding material will be polymerized for 60 seconds for each block after trays removal. At the end of the polymerization process, the blue bonding material excess will be removed with white stone finishing bur.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age (8-11) years (CVM stages 2-3)
* Mild class III skeletal pattern (Wits appraisal = 0 to -8)
* Mixed dentition
* Mild to moderate reverse overjet (-1 to -4)
* Overbite (1-5)
* Average or below average maxillary mandibular plane angle and lower facial height
* Mild incisors compensations

Exclusion Criteria:

* Severe class III skeletal pattern
* Long facial height
* Bad oral hygiene
* Systemic condition that may interfere with treatment
* No premolars or deciduous molars

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Dentoalveolar and skeletal effect of Digital bonded Reverse Twin Block in mixed dentition | 12 months
  Digital Bonded Reverse Twin Block is composed of four fixed blocks , 2 blocks cemented on upper premolars or deciduous molars & 2 blocks cemented on lower permanent molars with inclined planes 70 degrees One of the most engaging aspects of the DBRTB is its immediate facial treatment effects. Patient and their parents, immediately had the perception of facial profile modification. These facial changes can significantly improve the psychological patient's condition, improving their self-esteem and potentially making patients more confident.
  The digital workflow allows full appliance customization creating a perfect adaptation of the four blocks with patient dental anatomy thus optimizing bonding procedures and block retention.
  The dental effect of DBRTB is proclination of upper incisors, retroclination of lower incisors The skeletal effect of DBRTB is evaluated from cephalometric measurements: increase in SNA, decrease in SNB and ANB after ttt of mild skeletal class III cases
Dentoalveolar and skeletal effect of Digital bonded Reverse Twin Block in mixed dentition | 12 months
  Digital Bonded Reverse Twin Block is composed of four fixed blocks , 2 blocks cemented on upper premolars or deciduous molars & 2 blocks cemented on lower permanent molars with inclined planes 70 degrees.
  One of the most engaging aspects of the DBRTB is its immediate facial treatment effects. Patient and their parents, immediately had the perception of facial profile modification. These facial changes can significantly improve the psychological patient's condition, improving their self-esteem and potentially making patients more confident.
  The digital workflow allows full appliance customization creating a perfect adaptation of the four blocks with patient dental anatomy thus optimizing bonding procedures and block retention.
  The dental effect of DBRTB is proclination of upper incisors, retroclination of lower incisors The skeletal effect of DBRTB is evaluated from cephalometric measurements: increase in SNA, decrease in SNB and ANB after ttt of mild skeletal class III cases

SECONDARY OUTCOMES:
OHRQoL (Oral Health-related Quality of Life) assessments are being incorporated into clinical studies and trials to measure efficaciousness of treatment with the goal of improving care. | 12 months
  Studies involving OHRQoL seek to measure changes in scores from baseline to post-treatment.
  The greater the malocclusion (skeletal class III), the lower the QoL. Researchers studying oral health problems have used OHRQoL as an outcome measure to determine the effect of treatment on QoL.
  The use of OHRQoL as an evaluative outcome measure is congruent with patient-centered care. Along with other clinical assessments, it allows oral healthcare professionals to evaluate the efficacy of treatment protocols from patients' perspectives.
  OHRAoL accurately weighs the risks and benefits associated with treatment. In addition, it provides evidence that costs associated with treatment protocols are worth the expense if they generally improve patients' OHRQoL we should consider sociocultural and psychological factors when assessing needs, outcomes, and clinical practice.
  A final consideration in the use of OHRQoL as an outcome measure is addressing and measuring clinically meaningful change.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt